CLINICAL TRIAL: NCT05567211
Title: Prevention of Energy Deficit Syndrome in Female Athletes. Molecular Mechanisms Associated With Malnutrition: Oxidative Stress and Other Physiological, Physical and Psychological Alterations.
Brief Title: Prevention of Energy Deficit Syndrome in Female Athletes. Molecular Mechanisms Associated With Malnutrition.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alicante (Other)
Responsible Party: Principal Investigator, Prof. Dr. Alejandro Martínez-Rodríguez, Full Professor, University of Alicante
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UA-2021-03-11
Record Dates: First submitted 2022-09-30; First posted 2022-10-05 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Female Athlete Triad; Energy Deficit Syndrome; Mediterranean Diet; Red Fruits; Antioxidative Stress; Nutritional Disorder; Sports Physical Therapy
MeSH Terms: conditions — Female Athlete Triad Syndrome; Nutrition Disorders | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (No Intervention): Will receive basic recommendations from the World Health Organization on healthy eating and physical activity.
- Control group with free use of the virtual platform (Placebo Comparator): The athletes, in addition to the recommendations indicated in the previous point, will have access to the virtual platform designed to voluntarily record the parameters they consider appropriate.
  Interventions: Other: Free use of the virtual platform.
- Intervention group with Mediterranean diet and physical exercise planning (Active Comparator): They will receive nutritional plans adapted to their energy expenditure and based on Mediterranean diet. The physical exercise intervention will be based on 3 weekly sessions of 50 minutes of combined resistance and strength, deferred.
  Interventions: Other: Personalized nutritional planning based on the Mediterranean diet + physical exercise + use of mobile application.
- Intervention group with red berries and physical exercise planning (Active Comparator): They will also receive personalized nutritional plans with a diet rich in antioxidants obtained from red berries and the same physical exercise intervention as in the Mediterranean diet intervention group.
  Interventions: Other: Personalized nutritional planning with an extra intake of berries + physical exercise + use of mobile application.

INTERVENTIONS:
Other: Free use of the virtual platform. — Access to the virtual platform + general healthy eating and physical activity recommendations. The platform will allow the registration of all the evolution, monitoring of nutritional and sports patterns (with activity bracelet), as well as oxidative stress, hydration, menstrual phase and mood.
  Arms: Control group with free use of the virtual platform
Other: Personalized nutritional planning based on the Mediterranean diet + physical exercise + use of mobile application. — Access to the virtual platform + nutritional planning based on the Mediterranean diet + physical activity. The platform will allow the registration of all the evolution, monitoring of nutritional and sports patterns (with activity bracelet), as well as oxidative stress, hydration, menstrual phase and mood.
  Arms: Intervention group with Mediterranean diet and physical exercise planning
Other: Personalized nutritional planning with an extra intake of berries + physical exercise + use of mobile application. — Access to the virtual platform + nutritional planning with an extra supply of antioxidants using red berries + physical activity. The platform will allow the registration of all the evolution, monitoring of nutritional and sports patterns (with activity bracelet), as well as oxidative stress, hydration, menstrual phase and mood.
  Arms: Intervention group with red berries and physical exercise planning

SUMMARY:
Energy Deficit Syndrome (RED-S) is the impairment of physiological functioning caused by relative energy deficiency and includes impaired metabolic rate, menstrual, endocrine, hematological, immunological, gastrointestinal, bone, psychological, developmental and cardiovascular function. Eighty-seven percent of athletes show at least one symptom related to RED-S, with a higher prevalence in women. Treatment of RED-S preferably involves a multidisciplinary team of health professionals to address the complex interaction of nutrition, training, body image and performance. The main objective is to prevent energy deficit syndrome in female athletes in the province of Alicante through different training and diet protocols using a virtual platform. A 12-week single-blind randomized clinical trial with an intervention period and a control period (RCT) is proposed. The sports federations of the most representative practices in the province of Alicante will be selected by randomized sampling. The female athletes will be randomly divided into 4 groups (control group; control group with free use of the virtual platform; intervention group with Mediterranean diet and physical exercise planning; intervention group with red fruits and physical exercise planning).

ELIGIBILITY:
Inclusion Criteria:

* (a) exercise at least 3 days/week,
* (b) not having any diagnosed chronic pathology or ailment that prevents physical exercise or following nutritional guidelines rich in antioxidants.

Exclusion Criteria:

- All individuals taking medication that could affect the results of the study will be excluded from the study.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Oxidative stress | 12 weeks
  Measurement of oxidative stress by pentane by exhaled air
Weight | 12 weeks
  Weight evaluation using a digital scale
Anthropometric assessment - Height | 12 weeks
  Restricted profile proposed by the International Society for the Development of Cineanthropometry.
Fat mass | 12 weeks
  Through anthropometry. Restricted profile proposed by the International Society for the Development of Cineanthropometry. The Faulkner formula will be used.
Muscular mass | 12 weeks
  Through anthropometry. Restricted profile proposed by the International Society for the Development of Cineanthropometry. Lee's formula will be used.
Bone mass | 12 weeks
  Through anthropometry. Restricted profile proposed by the International Society for the Development of Cineanthropometry. The Rocha formula will be used.
Hydratation | 12 weeks
  Urine density will be measured with Refractometer.
Menstrual cycle | 12 weeks
  Using the Relative Energy Deficiency in Sport (RED-S) Clinical Assessment Tool (CAT) questionnaire. It is a clinical assessment tool for the evaluation of athletes / active individuals suspected of having relative energy deficiency and for guiding return to play decisions.
Gastrointestinal symptoms | 12 weeks
  The questionnaire on irritable bowel syndrome and symptom management among endurance athletes will be used; https://pubmed.ncbi.nlm.nih.gov/30232638/
Maximal oxygen uptake (VO2 max.) | 12 weeks
  In cycloergometer and cardiorespiratory fitness test monitored with electrocardiogram
Blood pressure | 12 weeks
  Using an OMROM upper arm blood pressure monitor.
Cholesterol in blood | 12 weeks
  Cholesterol by blood test
Strength | 12 weeks
  All participants will perform a countermovement jump, using a contact platform. Higher values will mean better performance.
Creatin-Kinase in blood | 12 weeks
  Creatin-Kinase by blood test (milligrams/deciliters). High values may be a sign of overtraining.
Perception of quality of life | 12 weeks
  Using a Quality of Life Questionnaire (SF36). Quality of Life Questionnaire is a comprehensive questionnaire that covers various attributes of an individuals life. It covers a variety of demographic questions to get better quality data and information before analyzing the quality of life of an individual.The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
Mood state | 12 weeks
  Profile of Mood State Questionnaire (POMS). The POMS questionnaire assesses six mood subscales: tension-anxiety, depression, anger-hostility, vigor, fatigue, and confusion. High vigor scores reflect a good mood or emotion, and low scores in the other subscales reflect a good mood or emotion.
Eating behavior | 12 weeks
  Eating Behavior Questionnaire (EAT-26). It is used to identify the presence of "eating disorder risk" based on attitudes, feelings and behaviours related to eating. There are 26 self-report questions assessing general eating behaviour and five additional questions assessing risky behaviours. The total score (between 0 and 78) provides an overall risk score, where higher scores indicating greater risk of an eating disorder. Total scores 20 or above are considered to be in the clinical range.

CONTACTS AND LOCATIONS:
Locations (1):
- Alejandro Martínez Rodriguez, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No